CLINICAL TRIAL: NCT05820763
Title: A Phase II Study of Selinexor In Addition to Lenalidomide for Consolidation and Maintenance Treatment After Autologous Hematopoietic Cell Transplant in Multiple Myeloma
Brief Title: Selinexor and Lenalidomide for Consolidation and Maintenance Treatment in Multiple Myeloma Post-transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study sponsor decided to close study.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202306068
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Myeloma-Associated Amyloidosis
Keywords: symptomatic multiple myeloma; myeloma post-AHCT; myeloma post-transplant; Multiple myeloma with amyloid deposition; Multiple Myeloma; post-transplant maintenance; Minimal residual disease
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — selinexor; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Patients will initially receive 4 cycles of consolidation triplet therapy followed by 8 cycles of maintenance doublet therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Consolidation: Selinexor, Lenalidomide, and Dexamethasone (Experimental): Consolidation will begin between Days 80 and 140 following standard of care autologous hematopoietic stem cell transplant and the treatment will consist of selinexor, lenalidomide, and dexamethasone for 4 28-day cycles.
  Interventions: Drug: Selinexor; Drug: Lenalidomide; Drug: Dexamethasone
- Maintenance: Selinexor and Lenalidomide (Experimental): Maintenance will consist of selinexor and lenalidomide for a maximum of 8 28-day cycles.
  Interventions: Drug: Selinexor; Drug: Lenalidomide

INTERVENTIONS:
Drug: Selinexor — Selinexor is administered by mouth on Days 1, 8, 15, and 22 at a dose of 60 mg during the four cycles of consolidation. Selinexor is then decreased to 40 mg and administered by mouth on Days 1, 8, 15, and 22 for up to 8 cycles of maintenance therapy.
  Other Names: EXPOVIO; KPT-330
Drug: Lenalidomide — Lenalidomide is administered by mouth daily on Days 1 to 21 at a dose of 10 mg during the first three cycles of consolidation, and then titrated up to 15 mg on Days 1 to 21 for the fourth cycle of consolidation. Lenalidomide 15 mg by mouth daily on Days 1 to 21 can be continued for up to 8 cycles of maintenance therapy.
  For patients with baseline renal dysfunction, the starting dose of lenalidomide will be 2.5 mg or 5 mg by mouth daily on Days 1 to 21. Patients may titrate up per physician discretion.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone is administered by mouth on Days 1, 8, 15, and 22 at a dose of 20 mg during all four cycles of consolidation only.
  Other Names: Decadron
  Arms: Consolidation: Selinexor, Lenalidomide, and Dexamethasone

SUMMARY:
This phase II clinical trial studies the addition of selinexor to lenalidomide in patients with multiple myeloma following transplant. Selinexor is an oral medication approved for use in patients with multiple myeloma following failure of other regimens, and lenalidomide is an oral medication approved for use in patients with multiple myeloma following transplant. This study is testing if the combination of selinexor and lenalidomide is more effective than lenalidomide alone in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age at time of enrollment.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Histologically confirmed diagnosis of multiple myeloma that is symptomatic. Patients with multiple myeloma with local amyloid deposition in the bone marrow are eligible.
* Patients must have undergone lenalidomide-based induction regimen.
* Patient must have undergone AHCT within 80 to 140 days prior to C1D1 for MM.
* Patient must be MRD-positive (per 10^-5 threshold) using clonoSEQ MRD® assay on bone marrow biopsy prior to study enrollment.
* Patient must have achieved very good partial response or better per IMWG response criteria prior to study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
* Adequate organ function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 K/cumm.
  * Platelet count ≥ 100 K/cumm (patients for whom <50% of bone marrow nucleated cells are plasma cells) or ≥50 K/cumm (patients for whom ≥50% of bone marrow nucleated cells are plasma cells).; platelet transfusions to help patients meet eligibility criteria are not allowed within 7 days before C1D1.
  * Hemoglobin ≥ 8.5 g/dL without blood transfusion within 7 days before C1D1.
  * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN), patients with Gilbert's syndrome must have a total bilirubin of < 3 x ULN.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN.
  * Calculated creatinine clearance ≥ 15 mL/min per Cockcroft and Gault formula.
* Women of childbearing potential must follow pregnancy testing requirements as outlined in the Revlimid REMS® program material. This is defined as either committing to continued abstinence from heterosexual intercourse or beginning TWO acceptable methods of contraception (one highly effective method and one additional effective method AT THE SAME TIME) at least 28 days prior to the start of lenalidomide, for the duration of study participation, and for 28 days following the last dose of lenalidomide. Women of childbearing potential must also agree to ongoing pregnancy testing.
* Men must agree to use a latex condom during sexual contact with a woman of childbearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* All study participants must be registered into the mandatory Revlimid REMS® program and be willing to comply with its requirements. Per standard Revlimid REMS® program requirements, all physicians who prescribe lenalidomide for research subjects enrolled into this trial, must be registered in, and must comply with, all requirements of the Revlimid REMS® program.

Exclusion Criteria:

* Patients with lenalidomide-refractory disease during induction.
* Prior receipt of selinexor or another XPO1 inhibitor previously.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Evidence of MM disease progression any time prior to enrollment. Progression from smoldering/asymptomatic MM to symptomatic MM is not exclusionary.
* Tandem autologous transplantation.
* History of plasma cell leukemia or MM CNS involvement.
* Administration or planned administration of any other concomitant chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy which would be considered a treatment of multiple myeloma from Day +28 post-transplant through discontinuation from study. Patients may be on corticosteroids if they are being given for disorders other than multiple myeloma (e.g., adrenal insufficiency, rheumatoid arthritis, etc.).
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Prior organ transplant requiring immunosuppressive therapy.
* Subjects with active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 IU/ml prior to first dose of trial treatment. Subjects with untreated hepatitis C virus (HCV) are allowed. Subjects with Human Immunodeficiency Virus (HIV) who have CD4+ T-cell counts ≥ 350 cells/µL and no history of AIDS-defining opportunistic infections in the last year are allowed.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
* Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
* Concurrent hematologic or non-hematologic malignancy requiring treatment (other than multiple myeloma with local amyloid deposition in the bone marrow).
* Active, unstable cardiovascular function, as indicated by the presence of:

  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (e.g. patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
  * Congestive heart failure of NYHA Class ≥3 or known left ventricular ejection fraction of <40%, or
  * Myocardial infarction within 3 months prior to C1D1.
* Grade > 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Major surgery within 14 days prior to C1D1.
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to C1D1. Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days prior to C1D1 and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Minimal Residual Disease (MRD) negativity | At the end of consolidation treatment (at the end of 4 cycles (each cycle is 28 days)
  Defined by rate of MRD negativity using clonoSEQ MRD® assay at a sensitivity of 10^-5. MRD negativity is defined as 0 residual clonal cells in a bone marrow biopsy sample.
Rate of Minimal Residual Disease (MRD) negativity | 12 months from study treatment initiation
  Defined by rate of MRD negativity using clonoSEQ MRD® assay at a sensitivity of 10^-5. MRD negativity is defined as 0 residual clonal cells in a bone marrow biopsy sample.

SECONDARY OUTCOMES:
Rate of partial response or better | 12 months from study treatment initiation
  Defined as the rate of patients achieving a partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR), as defined by standard IMWG response criteria.
Progression-free survival (PFS) | 12 months from study treatment initiation
  PFS will be defined as time from AHCT to progression, relapse, or death, whichever occurs first, and those event-free survivors will be censored at withdrawal or study closeout

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schroeder, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data underlying the results of the publication will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available immediately following publication, no end date.
Access Criteria: Researchers who provide a methodologically sound proposal for any purpose may request data. Proposal should be directed to markschroeder@wustl.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu